CLINICAL TRIAL: NCT01594398
Title: A Phase I Study to Assess the Food Effect on the Pharmacokinetics of Entinostat in Postmenopausal Women With Locally Recurrent or Metastatic ER+ Breast Cancer and Men and Women With Progressive Non-Small Cell Lung Cancer
Brief Title: Study to Assess Food Effect on Pharmacokinetics of Entinostat in Subjects With Breast Cancer or Non-Small Cell Lung Cancer
Acronym: ENCORE110
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Syndax Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SNDX-275-0110
Record Dates: First submitted 2012-05-04; First posted 2012-05-09 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Lung Cancer; Non Small Cell Lung Cancer (NSCLC); Breast Cancer; Estrogen Receptor Breast Cancer
Keywords: carcinoma,non small cell lung; lung diseases; lung neoplasms; Respiratory; Carcinoma, Bronchogenic; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Respiratory Tract Diseases; Erlotinib; Protein Kinase Inhibitors; Breast Neoplasms; Neoplasms; Breast Diseases; Exemestane; Aromatase Inhibitors
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Lung Diseases; Carcinoma, Bronchogenic; Bronchial Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Respiratory Tract Diseases; Neoplasms; Breast Diseases | interventions — entinostat; Erlotinib Hydrochloride; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- entinostat C1D1 fed (Experimental): Entinostat: Beginning C1D1 fed; C1D15 fasted. Erlotinib: NSCLC pts beginning C2D1,150 mg, po, qd. Exemestane: Breast cancer pts beginning C2D1,25 mg, po, qd.
  Interventions: Drug: entinostat; Drug: Erlotinib; Drug: Exemestane
- entinostat C1D1 fasted (Experimental): Entinostat: Beginning C1D1 fasted; C1D15 fed. Erlotinib: NSCLC pts beginning C2D1,150 mg, po, qd. Exemestane: Breast cancer pts beginning C2D1,25 mg, po, qd.
  Interventions: Drug: entinostat; Drug: Erlotinib; Drug: Exemestane

INTERVENTIONS:
Drug: entinostat — 10 mg, po, q14 days, until progression or intolerable toxicity
  Other Names: SNDX-275, MS-275
  Arms: entinostat C1D1 fed
Drug: entinostat — 10 mg, po, q14 days, until progression or intolerable toxicity
  Other Names: SNDX-275, MS-275
  Arms: entinostat C1D1 fasted
Drug: Erlotinib — Erlotinib: NSCLC pts beginning C2D1,150 mg, po, qd.
  Other Names: Tarceva
  Arms: entinostat C1D1 fed
Drug: Erlotinib — Erlotinib: NSCLC pts beginning C2D1,150 mg, po, qd.
  Other Names: Tarceva
  Arms: entinostat C1D1 fasted
Drug: Exemestane — Exemestane: Breast cancer pts beginning C2D1,25 mg, po, qd.
  Other Names: Aromasin
  Arms: entinostat C1D1 fed
Drug: Exemestane — Exemestane: Breast cancer pts beginning C2D1,25 mg, po, qd.
  Other Names: Aromasin
  Arms: entinostat C1D1 fasted

SUMMARY:
The purpose of this study is to evaluate the effect of food on the pharmacokinetics (PK) of the experimental drug, entinostat, in women with breast cancer and men and women with non-small cell lung cancer. The safety and tolerability of entinostat will also be evaluated when entinostat is given by itself as well as with the approved drugs, exemestane (Aromasin®) or erlotinib (Tarceva®). A biomarker (chemical "marker" in the blood/tissue that may be related to your response to the study drug) will also be tested.

DETAILED DESCRIPTION:
This is Phase 1, randomized, open-label, study of entinostat. The study is designed to evaluate any food effect on the pharmacokinetics of entinostat.

Patients will be randomized to receive entinostat with or without food on Cycle 1 Day 1 (C1D1). Patients randomized to receive entinostat with food on C1D1 will receive a second dose of entinostat without food on Cycle 1 Day 15 (C1D15). Patients randomized to receive entinostat without food on C1D1 will receive a second dose of entinostat with food on C1D15. Each cycle in the study will be for 28 days duration. Blood samples will be obtained pre-dose and serial blood samples will be taken after each dose to assess pharmacokinetics. For Cycle 2 and all subsequent cycles, all patients will continue to receive entinostat on Days 1 and 15 of each cycle. Those with breast cancer will also receive exemestane orally once daily starting on Cycle 2 Day 1. Those with NSCLC will also receive erlotinib starting on Cycle 2 Day 1.

Patients will be assessed at screening and at pre-prescribed times during study enrollment using standard assessments. Patients will also be assessed for tumor response after each 2 cycles. Patients will continue receiving study treatment until tumor progression or adverse events occur which necessitate discontinuing therapy as determined by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

Breast Cancer Patients Only

* Postmenopausal female patients
* Histologically or cytologically confirmed ER+ breast cancer at initial diagnosis and now has current disease progression and is a candidate to receive exemestane

NSCLC Patients Only:

* Cytologically or histologically confirmed NSCLC of stage IIIb or IV
* Received 1 to 2 prior chemotherapy or chemoradiotherapy regimens for advanced NSCLC (excluding erlotinib and valproic acid) and now has disease progression and is a candidate to receive erlotinib

All Patients:

* Age ≥ 18 years
* Patient must have the following laboratory parameters at study screening: Hemoglobin ≥ 9.0 g/dL; unsupported platelets ≥ 100.0 10-9/L; ANC ≥ 2.0 x 10-9/L; Creatinine less than 2.5 times the upper limit of normal for the institution; AST and alanine transaminase (ALT) < 2.5 times the upper limit of normal for the institution
* Patients may have a history of brain metastasis as long as certain criteria are met

Exclusion Criteria:

* Pregnant or lactating women
* Patient has rapidly progressive or life-threatening metastases.
* Patient has had previous treatment with entinostat or any other HDAC inhibitor including valproic acid
* Patient has a concomitant medical condition that precludes adequate study treatment compliance or assessment, or increases patient risk in the opinion of the investigator, such as but not limited to:

MI or arterial thromboembolic events within 6 months, or experiencing severe or unstable angina, New York Heart Association (NYHA) Class III or IV disease and a QTc interval > 0.47 seconds.

Uncontrolled heart failure or hypertension, uncontrolled diabetes mellitus, uncontrolled systemic infection.

* Patients with another active cancer (excluding adequately treated basal cell carcinoma or cervical intraepithelial neoplasia [CIN / cervical carcinoma in situ] or melanoma in situ). Prior history of other cancer is allowed, as long as there is no active disease within the prior 5 years.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Difference in pharmacokinetics of entinostat when subjects fed or fasted | C1D1 (sequential), D2, 4, 6, 8, 11; C1D15 (sequential), 16, 18, 20, 22 25; C2D1
  The pharmacokinetics of entinostat will be analyzed from patient plasma samples: maximum plasma concentration, time of maximum plasma concentration, area under the plasma concentration-time curve from baseline to last measurable concentration and extrapolated to infinity, terminal elimination rate constant.

SECONDARY OUTCOMES:
Change in laboratory values from baseline | Screening, C1D1, C1D15, C2D1, C3D1
  Chemistry, hematology blood samples: changes from baseline will be evaluated.
Change in ECG results from baseline | Screening, C1D1 (sequential), D2, 4, 6, 8, 11; C1D15 (sequential), D16, 18, 20, 22, 25; C2D1; EOT
  Changes from baseline will be evaluated including analysis of QTc prolongation and QTc change from baseline.
Difference in pharmacodynamics from baseline | C1D1, D2, D8; C1D15, D16, D22; C2D1; C3D1; EOT
  Blood samples will be analyzed for changes from baseline in protein lysine acetylation as measured by peripheral blood monocytes. The food effect, changes after entinostat, and changes after exemestane and erlotinib will be evaluated.
Adverse events | C1D1 , D2, 4, 6, 8, 11; C1D15, 16, 18, 20, 22 25; C2D1; D1 of each subsequent cycle through end of treatment
  Incidence of treatment emergent adverse events, serious adverse events, adverse events resulting in permanent discontinuation of study drug, and deaths occurring within 30-days of the last dose of study drug.

CONTACTS AND LOCATIONS:
Overall Officials: William McCulloch, M.D., Study Director — Syndax Pharmaceuticals; Howard A Burris, M.D., Principal Investigator — Tennessee Oncology
Locations (3):
- United States (3):
  - Florida Cancer Specialists, Sarasota, Florida
  - Peggy and Charles Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Sarah Cannon Research Institute, Nashville, Tennessee

REFERENCES:
- [Background] Witta SE, Jotte RM, Konduri K, Neubauer MA, Spira AI, Ruxer RL, Varella-Garcia M, Bunn PA Jr, Hirsch FR. Randomized phase II trial of erlotinib with and without entinostat in patients with advanced non-small-cell lung cancer who progressed on prior chemotherapy. J Clin Oncol. 2012 Jun 20;30(18):2248-55. doi: 10.1200/JCO.2011.38.9411. Epub 2012 Apr 16. PMID 22508830